CLINICAL TRIAL: NCT06069791
Title: Anesthetic Greater Occipital Nerve Blockade in Veterans With Post-Traumatic Headache: Sub-study 1
Brief Title: Greater Occipital Nerve Blockade in Veterans With Post-concussion Headache: Sub-study 1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Headache Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1656679
Record Dates: First submitted 2023-09-28; First posted 2023-10-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Post-Traumatic Headache
Keywords: traumatic brain injury; veteran; VA Connecticut Healthcare System
MeSH Terms: conditions — Post-Traumatic Headache; Brain Injuries, Traumatic | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: incomplete block assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both bupivacaine concentration and order of administration will be unknown except to Research Pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): bupivacaine 0.0%, 0.01%, and 0.05% in random order, one week apart each
  Interventions: Drug: Bupivacaine Injection
- Group 2 (Experimental): bupivacaine 0.1%, 0.05%, and 0.1% in random order, one week apart each
  Interventions: Drug: Bupivacaine Injection
- Group 3 (Experimental): bupivacaine 0.0%, 0.1%, and 0.5% in random order, one week apart each
  Interventions: Drug: Bupivacaine Injection
- Group 4 (Experimental): bupivacaine [0.01% or 0.05%], [0.05% or 0.1%], and 0.05% in random order, one week apart each
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — subcutaneous injection around bilateral greater occipital nerves

SUMMARY:
The acute and subacute sensations that occur on the scalp with injection of different concentrations of bupivacaine for grater occipital nerve blockade will be compared. Each Veteran participant will be randomized to receive three different concentrations, which will be injected one week apart each.

DETAILED DESCRIPTION:
Military Servicemembers are at elevated risk for traumatic brain injury (TBI) and its consequences, including post-traumatic headache (PTH). The most common phenotype of PTH is migraine, for which there are numerous potential treatments, though these have limitations, including poor efficacy, drug-drug interactions, and intolerable side effects. Therefore, the consideration of other methods to manage PTH in Servicemembers and Veterans is warranted.

Anesthetic greater occipital nerve (GON) blockade is a simple, inexpensive, and safe procedure that has demonstrable headache pain suppressing effects in a variety of headache disorders. This intervention is frequently done to provide immediate relief, followed by a period of reduced headache burden.

The acute burning that occurs during injection and then the numbing over the scalp that occurs shortly after anesthetic GON blockade make controlled investigations against placebo difficult to interpret. In sub-study 1 of this project, different concentrations of bupivacaine (0.0%, 0.01%, 0.05%, 0.1%) will be examined in order to identify a suitable control dose to later compare to the full dose of 0.5%. Acute and subacute sensations from bupivacaine GON blockade will be measured and the lowest concentration that resembles the sensations elicited by full dose (0.5%) will be used in a subsequent efficacy trial (sub-study 2).

ELIGIBILITY:
Inclusion Criteria:

* United States Military Veterans within VA Connecticut Healthcare System
* Chronic post-traumatic headache per ICHD-3 criteria (i.e., headaches are continuing to occur three months after the head injury)
* At least two headache days per week
* MRI brain scan completed within the past 3 months if chronic PTH for less than one year, within the past year if chronic PTH for less than 5 years, and within 5 years if chronic PTH for more than 10 years
* Review of MRI and the medical record does not reveal another source for headache

Exclusion Criteria:

* Skull defect
* Other contraindication to bupivacaine

  1. Allergy or adverse reaction (e.g., rash, cardiac effects) to amide anesthetics, such as lidocaine
  2. Instruction from clinician to avoid amide anesthetics, such as lidocaine
* Pregnant or lack of adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute sensation felt during injection: quality | During injection
  The quality of the sensation on the scalp at the time of injection (e.g., burning, shooting, aching)
Acute sensation felt during injection: intensity | During injection
  The maximum intensity of the sensation on the scalp at the time of injection on 0-10 numerical rating scale
Paresthesia felt after injection: quality | From the time of injection to 1 week after injection
  The quality of the sensation over the scalp after injection (e.g., numbing, tingling, coolness)
Paresthesia felt after injection: intensity | From the time of injection to 1 week after injection
  The maximum intensity of the sensation over the scalp after injection on 0-10 numerical rating scale
Paresthesia felt after injection: distribution | From the time of injection to 1 week after injection
  The location of the sensation over the scalp after injection, drawn on figure of head and neck
Paresthesia felt after injection: duration | From the time of injection to 1 week after injection
  The duration of the sensation over the scalp after injection (hours)

SECONDARY OUTCOMES:
Adverse events | From the first injection to two weeks after the last injection
  Complications that occur during or after injection

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No